CLINICAL TRIAL: NCT06575465
Title: Examining the Effectiveness of Family and Community-Based Intervention Programs to Improve Treatment Adherence for Overweight, Obesity, Prediabetes, Metabolic Syndrome, and Type 2 Diabetes in the Bedouin Community in the Negev
Brief Title: Evaluating Family & Community-Based Interventions to Improve Treatment Adherence in Metabolic Health Among Negev Bedouins (EFIT-BED)
Acronym: EFIT-BED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Vered Kaufman Shriqui, Associate Professor, Ariel University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0133-23-COM
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Community-Based Participatory Research
Keywords: Type 2 Diabetes Mellitus; Obesity; Community based participatory research; Health promotion; Clinical trial; Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Prediabetic State | interventions — Culture Techniques

STUDY DESIGN:
Intervention Model Description: Study Design: The study is designed as a controlled community intervention trial. Participants will be divided into two groups: an intervention group and a control group. The intervention group will receive a comprehensive community-based intervention program, while the control group will receive routine care.
  Intervention Group:
  * Will receive a tailored healthy lifestyle intervention program focusing on nutrition, physical activity, and behavioral changes.
  * 10 sessions will be conducted separately for men and women.
  * Each session will last for approximately 2 hours.
  * The program will include educational workshops, cooking demonstrations, physical activity sessions, and group discussions.
  Control Group:
  • They will continue to receive standard care from their healthcare providers without additional intervention.
  Duration of the Study:
  • The study will last for one year, with follow-up assessments conducted at baseline, 6 months, and 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full Intervention (Experimental): * Will receive a tailored healthy lifestyle intervention program focusing on nutrition, physical activity, and behavioral changes.
  * Ten sessions will be conducted separately for men and women.
  * Each session will last for approximately 2 hours.
  * The program will include educational workshops, cooking demonstrations, physical activity sessions, and group discussions.
  Interventions: Behavioral: Healthy lifestyle nutrition, culture and physical activity workshops
- Control group (Active Comparator): Participants will continue to receive standard care from their healthcare providers without additional intervention.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Healthy lifestyle nutrition, culture and physical activity workshops — The intervention will include monthly sessions in the community setting of physical activity. In addition, monthly nutrition and culture sessions will be held.
  Arms: Full Intervention
Other: Usual care — Usual care patients receive in their primary health care
  Arms: Control group

SUMMARY:
Background:

The Bedouin community in the Negev faces high rates of type 2 diabetes, low treatment adherence, and increased disease complications. Transition to urban living and changing dietary patterns have exacerbated these issues. Current interventions often overlook the potential of culturally tailored approaches leveraging kinship ties and community resources. This study seeks to address these gaps by examining the impact of a family-centered intervention program.

Objectives:

Primary: Assess the effect of community intervention on Mediterranean diet adherence.

Secondary: Evaluate changes in fasting glucose, HbA1c, lipid profiles, BMI, physical activity, and quality of life.

Methodology:

Study Design: Controlled community intervention trial with two groups (intervention and control).

Participants: 170 Bedouin adults diagnosed with overweight, obesity, metabolic syndrome, prediabetes, or type 2 diabetes.

Intervention: 10 sessions over 12 months focusing on nutrition, physical activity, and behavioral changes, tailored to cultural norms.

Control: Routine care without added intervention. Outcome Measures: Lab tests (HbA1c, lipid profiles), anthropometric measures, Mediterranean diet adherence, physical activity, quality of life, and social belonging.

Recruitment and Data Collection:

Participants will be recruited via Clalit clinics in Rahat, with the support of local community leaders. Data will be collected through medical records, questionnaires, and physical assessments at baseline, 6, and 12 months.

Data Analysis:

Statistical analysis will be performed using SAS/SPSS, employing ANOVA, Chi-square tests, and regression models for outcome prediction.

Ethical Considerations:

Participants' privacy will be ensured through coded data storage. The study will comply with Helsinki guidelines, and participants can withdraw at any time.

Conclusion:

This study aims to provide culturally tailored interventions to improve health outcomes in the Bedouin community, potentially serving as a model for similar minority groups globally.

DETAILED DESCRIPTION:
Research Initiator: Prof. Vered Kaufman-Shriqui, Department of Nutrition Sciences, Ariel University, Ariel. Email: veredks@ariel.ac.il Clalit HMO Principal Investigator: Dr. Muflah Ataika, Rahat Counseling Clinic, Southern District, Clalit Health Services.

Co-Investigators:

* Dr. Walid El Huzayel, Rahat A Clinic, Southern District, Clalit Health Services.
* Ms. Malak Oubra Abu Alasal, Regional Diabetes Nurse, Southern District, Clalit Health Services.

External Co-Investigators:

* Prof. Mona Boaz, Head of the Department of Nutrition Sciences at Ariel University in Samaria.
* Dr. Maya Maor, Department of Sociology and Anthropology, Ariel University.
* Dr. Samira Alfayoumi Ziadna, Ashkelon College.

Scientific Background and Rationale for the Study The health status of populations is shaped by social, political, economic, and cultural factors that influence individual behaviors. Social and cultural patterns are especially relevant in the context of diabetes, where lifestyle choices, diet, and physical activity play critical roles (Inoyue, 2012). A comprehensive approach targeting all sectors is essential for effective health promotion. However, despite widespread health initiatives, little is known about their long-term impact and sustainability.

The Bedouin community in the Negev has some of the highest rates of type 2 diabetes in Israel, with 40% of those over 50 affected (internal district data). Despite high disease prevalence, there are low success rates in disease management and high rates of complications. The Bedouin society is experiencing a cultural shift from a semi-nomadic lifestyle to permanent housing, which is altering traditional dietary habits (e.g., home-cooked meals vs. ready-made food). The extent to which these changes contribute to rising obesity and diabetes rates is unclear. Additionally, most research on diabetes in the Bedouin community focuses on adherence to standard interventions without considering how cultural norms could serve as unique coping resources (Maor et al., 2023). Studies on other minority groups suggest that community experiences and worldviews can enhance disease management strategies (Chard, 2017; Duwe, 2016; Sanderson, 2012).

Given the Bedouin society's strong clan ties, strategies involving collective actions (e.g., family-wide physical activities) may boost participation and treatment adherence (Maor et al., 2023). Therefore, tailored health promotion programs are essential for reducing health disparities in this community.

In Israel, despite overall high life expectancy, minority groups-especially those in lower socioeconomic strata-experience significantly shorter life spans. This gap is largely due to higher rates of chronic conditions like obesity and heart disease among Arab populations (Swinburn et al., 2011; ICDC, 2012). A 1999-2000 survey found that obesity rates (BMI > 30) in the Arab sector are notably high (Abdeen et al., 2012). A subsequent study involving 17,044 Arab participants (49% men; average age 39.4) and 16,012 Jewish participants (50% men; average age 40.5) confirmed significantly higher BMI and other risk factors (e.g., HDL-C, triglycerides, SBP) in the Arab population (Abdeen et al., 2012; Kalter-Leibovici et al., 2012).

The prevalence of type 2 diabetes in the Arab sector is roughly double that of the Jewish sector (Kalter-Leibovici et al., 2012; Abdeen et al., 2012). Adherence to treatment is particularly low among Bedouins, with over 70% of patients non-compliant, leading to severe complications such as kidney failure and blindness (Chard, 2017; Duwe, 2016). This highlights an urgent need to understand how Bedouin patients manage their condition.

Research Objectives General Objective: This study aims to evaluate whether a community-based intervention targeting healthy lifestyle practices within Bedouin clans can improve physical activity, glycemic control, anthropometric measures, and dietary habits in individuals with metabolic syndrome, prediabetes, and type 2 diabetes beyond routine medical care provided by physicians and clinic staff.

Primary Objective:

To examine the effect of the intervention on the Mediterranean diet score among patients with obesity, metabolic syndrome, prediabetes, and type 2 diabetes over a period of up to one year from their entry into the study.

Secondary Objectives: Among people with overweight, obesity, metabolic syndrome, prediabetes, and type 2 diabetes over a period of up to one year, to examine the effect of the community intervention on:

1. Fasting blood sugar levels (FPG) and glycosylated hemoglobin levels (HBA1c)
2. Blood lipid profile (LIPID PROFILE)
3. Anthropometric measures (weight, BODY MASS INDEX (BMI), waist circumference, blood pressure)
4. Nutritional intake quality
5. Health habits and physical activity level
6. Quality of life
7. Sense of social belonging We aim to examine whether a healthy lifestyle intervention program within the clan in the research group compared to the control group will lead to improvements in these outcome measures.

Number of Participants and Planned Study Centers:

Number of participants in the study: 170 participants Each intervention group requires 70 people (total 140 participants) + 15 participants in each group in case of dropout (total 170 participants). The intervention group will receive a program to promote a healthy lifestyle. The intervention will be given separately to men and women. There will be 10 meetings. The meeting topics are detailed in the research timeline table. The control group will not receive an intervention program.

The sample size was based on the following assumptions: The sample size was calculated to demonstrate a difference of 0.5±1% in HbA1c levels in a two-sided test α=0.05.

Participant Recruitment Method: Patients insured by Clalit Health Services from two selected clans in Rahat, whose elders agreed to participate in the study, from the Southern District, men and women aged 18 and above, will be recruited by the researchers in the study who are the primary treating physicians identifying suitable patients for participation in the study according to inclusion and exclusion criteria. Recruited patients will be referred for further testing and treatment.

Study Design and Methodology:

Study Design: The study is designed as a controlled community intervention trial. Participants will be divided into two groups: an intervention group and a control group. The intervention group will receive a comprehensive community-based intervention program, while the control group will receive routine care. All outcome measures will be measured at baseline, 6 months from baseline and 12 months from baseline.

Reporting of Adverse Events / Serious Adverse Events:

o At each visit, patients will be questioned about changes in their medical condition and changes in their regular medications. If an adverse event or serious adverse event occurs, it will be reported to the principal investigator and the study initiator according to the requirements of the Helsinki Committee and GCP procedures. The principal investigator will complete an Adverse Event or Serious Adverse Event report form as required.

* The principal investigator will compile data from all participating clinics.
* Each patient will be assigned a coded number in a sequential order, consisting of the initials of the patient's name and their recruitment order in the study. Identifying details will be omitted.
* The encrypted data file will be stored on the principal investigator's computer in the office of Dr. Muflah Ataika at the Clalit Health Services district management in Be'er Sheva.
* Study documents, including informed consent forms, research questionnaires, and other related materials, will be stored in a locked cabinet at the research site with restricted access to the research team only, according to good clinical practice (GCP) procedures.
* Identifying details will not be transferred to the study initiator outside of Clalit facilities; only coded data will be transferred.

Laboratory Tests and Any Other Relevant Tests to be Conducted During the Study and Follow-Up Period, and Where They Will Be Performed:

• Laboratory tests will not be specifically conducted for the study but will be extracted from the participants' medical records during each clinic visit. Anthropometric measurements will be actively checked at each meeting.

Method of Analyzing and Processing Results:

* Descriptive and inferential statistical analyses will be performed using SAS and/or SPSS software.
* For continuous variables, a normal distribution analysis will be conducted and, if necessary, a logarithmic transformation.
* Comparisons between continuous variables will be performed using appropriate statistical tests such as ANOVA (general comparison, and if necessary, between all groups and between each pair of groups).
* Comparisons of categorical variables will be performed using the Chi-square test and, if possible, the Fisher Exact test.
* For continuous outcome variables, a multivariate prediction model will be built, including demographic background factors of the participants and the intervention group they were part of.
* Multivariate comparisons will be conducted using logistic regression or multivariate linear regression as appropriate.

Role of the Sub-Investigators in the Study:

The sub-investigators will oversee all stages of the study implementation and intervention, including training research assistants on research questionnaires and medical teams (dietitians and physiotherapists) to integrate the intervention among the population. Additionally, they will supervise data collection, oversee the work of research assistants, conduct statistical analyses (on de-identified data), and write the research findings.

7. Ethical Issues of the Trial

* All subjects will sign an informed consent form prior to inclusion in the study.

  - Pregnant women, special populations, individuals lacking judgment capacity, and children will not be recruited for the study.
* Participants can withdraw from the study at any time.
* Number of centers in the study: This study involves one center, the primary investigator's clinic.

ELIGIBILITY:
Inclusion Criteria:

* Bedouin men and women aged 18 and above
* Diagnosed with overweight, obesity, metabolic syndrome, prediabetes, or type 2 diabetes
* Consent to participate in the study

Exclusion Criteria:

* Individuals with other chronic diseases that might interfere with the study
* Pregnant or lactating women
* Individuals unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of the intervention on the Mediterranean diet score among patients with obesity, metabolic syndrome, prediabetes, and type 2 diabetes over a period of up to one year from their entry into the study | Will be examined three times during one year
  Examine changes in Mediterranean score using the Mediterranean diet questionnaire (I-MEDAS), the score ranges from 0-17, with a higher value indicating better adherence to the Mediterranean diet pattern.

SECONDARY OUTCOMES:
Fasting blood sugar levels (FPG) | Three times during a year
  Level of fasting glucose
Levels of glycosylated hemoglobin levels (HBA1c) | Three times during a year
  Level of HBA1C
Blood lipid profile (LIPID PROFILE) | Three times a year
  Outcomes of a full lipid profile
Anthropometric measures (weight) | Three times during a year
  Weight will be measured in kilograms.
Anthropometric measures (waist circumference) | Three times during a year
  Waist circumference will be measured in centimeters.
Anthropometric measures (height) | Three times during a year
  Height will be measured in meters.
Body mass index, (BMI) | Three times during a year
  Weight and height will be combined to report BMI in kg/m^2
Blood pressure | Three times during a year
  Systolic and diastolic blood pressure in mm/Hg
Health habits and physical activity level | Three times during a year
  Assessed using a health and physical activity habits questionnaire. Smoking habits will be self reported.
Reported quality of life | Three times during a year
  Evaluated using the European Quality of life-5 Dimension (EQ-5D-5L) questionnaire measures health related quality of life. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state
Sense of belonging | Three times during a year
  Assessed using a social and community belonging questionnaire. The score ranges from 10-30, higher score indicates higher sense of belonging.

CONTACTS AND LOCATIONS:
Overall Officials: Muflah Ataika, MD, Principal Investigator — Rahat Counseling Clinic, Southern District, Clalit Health Services.
Locations (1):
- Clalit healthcare clinic, Rahat, Israel

IPD SHARING:
Plan to Share IPD: No